CLINICAL TRIAL: NCT05379959
Title: Effects of Stimulants on Behavioral and Neural Markers of Social Motivation, Ability, and Neural Markers of Social Function
Acronym: MASM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB21-1568
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Stimulant Use; MDMA ('Ecstasy'); Social Behavior; Motivation
MeSH Terms: conditions — Social Behavior | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Methamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental: Placebo Then MDMA Then Methamphetamine (Experimental): Participants first receive placebo at their first session in the laboratory. Then will return to the laboratory 5 days later and will receive 125 mg MDMA. Finally, 5 days later will return to the laboratory and will receive 20 mg of MA.
  Interventions: Drug: MDMA; Drug: Methamphetamine; Drug: placebo oral tablet
- Experimental: MDMA Then Placebo Then Methampetamine (Experimental): Participants first receive 125 mg of MDMA at their first session in the laboratory. Then will return to the laboratory 5 days later and will receive placebo. Finally, 5 days later will return to the laboratory and will receive 20 mg of MA.
  Interventions: Drug: MDMA; Drug: Methamphetamine; Drug: placebo oral tablet
- Experimental: Methampetamine Then Placebo Then MDMA (Experimental): Participants first receive 20 mg of MA at their first session in the laboratory. Then will return to the laboratory 5 days later and will receive placebo. Finally, 5 days later will return to the laboratory and will receive 125 mg of MDMA.
  Interventions: Drug: MDMA; Drug: Methamphetamine; Drug: placebo oral tablet

INTERVENTIONS:
Drug: MDMA — Participants will be given 125 mg of MDMA.
Drug: Methamphetamine — Participants will be given 20 mg of MA.
Drug: placebo oral tablet — Participants will be given a placebo capsule that will only contain lactose.

SUMMARY:
To study the effects of MDMA, compared to a prototypical stimulant, on social motivation, social ability, and neural indices of social function in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* BMI between 19 and 30 (no one under 130 lbs)
* Smokers smoking less than 25 cigarettes per week
* Have used ecstasy no more than 40 times with no adverse responses.

Exclusion Criteria:

* High blood pressure
* Any medical condition requiring regular medication
* Individuals with a current (within the last year) DSM-IV Axis 1 diagnosis
* Individuals with a history of dependence on stimulant drugs.
* Women who are pregnant or trying to become pregnant

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Profile of Mood States | Time Frame: Baseline-72 hours after completion of the sessions
  The POMS measures individuals' mood states. This is a validated scale to measure positive and negative mood states. The POMS contains 30 items and assesses six identified mood factors: Tension-Anxiety, Depression-Ejection, Anger- Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. Scoring of the instrument provides a global score of 0 to 120 or individual domain scores. Lower scores indicate better mood state. The POMS brief form is a simple self-rating instrument.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided